CLINICAL TRIAL: NCT07319429
Title: Refining Fertility-sparing Treatment in Endometrial Carcinoma Based on Molecular Classification: a Prospective Multicenter Umbrella Clinical Study（FEMUS）
Brief Title: Refining Fertility-sparing Treatment in Endometrial Carcinoma Based on Molecular Classification
Acronym: FEMUS
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Phd.MD. vice President, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20250520; SYYYRH2025010 (Other Grant/Funding Number: Shanghai Tenth People's Hospital)
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer; Fertility
Keywords: Fertility-sparing Treatment; Molecular Classification
MeSH Terms: conditions — Endometrial Neoplasms | interventions — spartalizumab; sintilimab; Medroxyprogesterone Acetate; Megestrol Acetate; Gonadotropin-Releasing Hormone; Letrozole

STUDY DESIGN:
Intervention Model Description: This is a non-randomized controlled, prospective, multi-center, umbrella clinical trial implementing stratified management based on molecular subtypes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- POLEmut Stage II Single-Arm Interventional Study (Experimental): Enroll patients with FIGO 2023 Stage IA POLE-mutant endometrial carcinoma to evaluate the CR rate, CR duration, and reproductive outcomes of ICI monotherapy in FST with expanded indications. Enrolled patients will receive ICI monotherapy.
  Interventions: Drug: PD1 antibody
- MMRd Stage II Single-Arm Interventional Study: (Experimental): Stratify patients based on MLH1 methylation status/MMR coding gene mutation status. Patients with MMR coding gene mutations (somatic/germline) will receive ICI monotherapy; MMRd patients with MLH1 promoter methylation will receive ICI combined with high-dose potent progestogens (PD-1 + MPA/MA). The study will evaluate the CR rate, CR duration, and reproductive outcomes of FST with expanded indications.
  Interventions: Drug: PD1 antibody; Drug: Medroxyprogesterone Acetate 500 MG; Drug: Megestrol Acetate 160 MG
- NSMP Stage III Two-Arm Interventional Study (Experimental): Based on the prediction model, progestogen-sensitive patients will receive high-dose potent progestogens (MA/MPA); progestogen-insensitive patients will receive "GnRHa combined with letrozole". The study will evaluate FST efficacy and reproductive outcomes while further validating the predictive value of the model.Exclusion from FST: NSMP EC with ER negativity and/or L1CAM positivity (≥10%) or p53abn endometrial carcinoma.
  Interventions: Drug: Medroxyprogesterone Acetate 500 MG; Drug: Megestrol Acetate 160 MG; Drug: GnRH agonist and Letrozole

INTERVENTIONS:
Drug: PD1 antibody — Administration: 200 mg via intravenous infusion, once every 3 weeks. After no lesions are detected in two consecutive pathological examinations, the patient enters the maintenance treatment phase. The maintenance treatment duration shall not exceed 6 months. During the maintenance period, 400 mg via intravenous infusion is administered once every 6 weeks, for 4 consecutive times.
  Other Names: Sintilimab Injection
  Arms: MMRd Stage II Single-Arm Interventional Study:; POLEmut Stage II Single-Arm Interventional Study
Drug: Medroxyprogesterone Acetate 500 MG — - Medroxyprogesterone Acetate: 500 mg, orally once daily, continuously.
  Arms: MMRd Stage II Single-Arm Interventional Study:; NSMP Stage III Two-Arm Interventional Study
Drug: Megestrol Acetate 160 MG — - Megestrol Acetate: 160 mg, orally once daily, continuously.
  Arms: MMRd Stage II Single-Arm Interventional Study:; NSMP Stage III Two-Arm Interventional Study
Drug: GnRH agonist and Letrozole — * Triptorelin Acetate for Injection (or similar drugs): 3.75 mg per vial, intramuscular injection once every 4 weeks as one treatment course.
  * Letrozole Tablets: 2.5 mg, orally once daily, continuously.
  In the clinical trial conducted at the same center, only the same drug from the same manufacturer shall be used as the trial medication.
  Arms: NSMP Stage III Two-Arm Interventional Study

SUMMARY:
Endometrial cancer (EC) stands among the most common gynecological malignancies in developed countries and regions, with a notable trend toward younger age at onset. Correspondingly, the demand for fertility-sparing treatment (FST) has been increasingly prominent among young EC patients. High-potency progestogens remain the sole therapeutic option recommended by international guidelines for this patient population; however, approximately 30% of patients exhibit no response to such treatment.

The concept of EC molecular subtyping, proposed by The Cancer Genome Atlas (TCGA) in 2013, has revolutionized the diagnosis and management of EC. EC subtypes with distinct molecular features demonstrate substantial differences in biological behaviors and responses to pharmacotherapeutic interventions. Nevertheless, the role of molecular subtyping in guiding FST decision-making-both in terms of its applicability and specific mechanisms-remains an unmet research need worldwide.

Notably, the POLE-mutant and microsatellite instability-high (MSI-H) subtypes display the highest sensitivity to immune checkpoint inhibitors, underscoring the clinical value of exploring their utility in FST. The no specific molecular profile (NSMP) subtype is sensitive to progestogens but lacks reliable predictive biomarkers-accurate pre-treatment prediction would enable tailored treatment selection, shorten treatment duration, and enhance therapeutic outcomes. In contrast, the p53-abnormal (p53abn) subtype is associated with a poor prognosis, and FST is therefore not recommended for this subgroup.

Building on the aforementioned background and our research team's preliminary clinical findings, this project focuses on the field of FST for EC. To address the current challenges-including narrow indications, limited treatment options, suboptimal efficacy, and the absence of precise personalized regimens-we aim to conduct the world's first prospective multicenter umbrella trial based on EC molecular subtyping. Optimal novel diagnostic and therapeutic protocols will be developed for each molecular subtype, with the goals of optimizing existing FST strategies, improving FST efficacy and reproductive outcomes, expanding eligible indications, and providing high-quality clinical evidence for molecular subtype-guided FST in EC, thereby advancing the overall effectiveness of FST for EC patients.

DETAILED DESCRIPTION:
1.Research Background Endometrial Carcinoma (EC) ranks among the most prevalent malignancies of the female reproductive system, with a globally increasing incidence and a notable trend toward younger age at onset, leading to a growing disease burden. Data from the U.S. National Cancer Institute indicates that the annual incidence of EC has increased by 1.5% over the past decade, with a particularly prominent rise among women under 50 years of age. The situation is equally severe in China: between 2004 and 2017, the crude incidence of EC rose from 6.20 to 10.06 per 100,000 population. In economically developed regions such as Beijing, Shanghai, and Tianjin, EC has become the most common gynecological malignancy. For Chinese women under 40, the crude incidence increased by 68.20% (from 0.63 to 1.07 per 100,000 in rural areas). This trend is closely associated with delayed childbearing, reduced parity, obesity, and the high prevalence of metabolic diseases like diabetes, predicting a continuous increase in EC-related burden over the next decade and highlighting the urgent need for systematic prevention and control strategies.

For young nulliparous EC patients, radical surgery-though the standard treatment-results in irreversible loss of fertility. Consequently, Fertility-Sparing Treatment (FST) has emerged as the core approach to balance tumor control and reproductive needs. However, FST for young EC patients currently faces critical bottlenecks:

1. Narrow indications and limited treatment options: Guidelines including NCCN， ESGO, and BGCS restrict FST eligibility to patients with well-differentiated (G1), FIGO 2009 Stage IA (confined to the endometrium) disease. Clinically, high-dose potent progestogens (medroxyprogesterone acetate [MPA], megestrol acetate [MA], and levonorgestrel-releasing intrauterine system [LNG-IUS]) remain the mainstay, yielding an overall complete response (CR) rate of only 70%-80%⁶.
2. Significant efficacy variability and prominent adverse effects: Even with our research team's modified regimen of "hysteroscopic lesion resection combined with high-dose progestogens"-which elevated the pathological CR rate to 97% (mean treatment duration: 6.42±0.45 months)-approximately 1/3 of patients require over 9 months of treatment or fail to achieve CR. Prolonged treatment not only increases the risk of endometrial damage due to repeated hysteroscopic evaluations and impairs ovarian function (affecting subsequent pregnancy) but also raises the risk of progestogen-related adverse events such as weight gain, liver dysfunction, thrombosis, and breast cancer. Concurrent symptoms including dizziness, headache, and gastrointestinal disturbances further reduce patients' quality of life and treatment adherence.
3. Lack of molecular subtype-guided precision protocols: The EC molecular classification system proposed by The Cancer Genome Atlas (TCGA) in 2013 (currently categorized into POLEmut, MMRd/MSI-H, NSMP, and p53abn subtypes) has revealed significant differences in biological characteristics and prognosis across subtypes (p53abn subtype has the poorest prognosis and is not suitable for FST; POLEmut subtype has the best prognosis; MMRd/MSI-H and NSMP subtypes have intermediate prognosis). While molecular subtyping has been incorporated into international guidelines such as ESGO/ESTRO/ESP¹¹ and ESMO to guide non-fertility-sparing EC management, research on subtype-specific personalized regimens, prediction of treatment non-responders, and alternative therapies in the FST setting remains severely insufficient, failing to meet clinical demands for precision medicine.

Advancements in EC molecular subtyping research and accumulating clinical evidence for immune checkpoint inhibitors (ICIs) have provided new opportunities to address these bottlenecks:

* POLEmut EC exhibits high tumor mutational burden (TMB-H) and robust immune responses, indicating significant potential for ICI treatment;
* Although MMRd/MSI-H EC shows poor response to progestogens, ICIs have demonstrated favorable efficacy in advanced and locally advanced cases;
* As the most common subtype, NSMP EC may benefit from progestogen therapy optimization through biomarker-based stratification.

Against this backdrop, conducting prospective clinical trials of molecular subtype-guided FST for EC has become an urgent priority to optimize FST strategies, improve therapeutic efficacy, and enhance reproductive and oncological outcomes.

2 Research Basis and Protocol Design for Each Molecular Subtype

1. POLEmut EC POLEmut EC accounts for approximately 10% of all EC cases, characterized by one of 11 pathogenic mutations in the POLE exonuclease domain (patients with non-pathogenic mutations have poorer prognosis), TMB-H, and dense tumor-infiltrating lymphocytes (TILs) with high PD-1 expression. Clinically, it exhibits excellent prognosis: the PORTEC-3 study showed that high-risk POLEmut EC patients achieved 5-year recurrence-free survival (RFS) rates of 100% and 97% with and without chemotherapy, respectively (p=0.64), and a 5-year overall survival (OS) rate of approximately 98%. The FIGO 2023 staging system classifies all uterine-confined POLEmut EC as Stage IA (Stage II patients are downgraded to Stage I for surveillance), and the RAINBO POLEmut-BLUE trial is currently exploring the feasibility of treatment de-escalation for this subtype.

   In the FST setting, hysteroscopic lesion resection remains the primary intervention, while systematic research on ICI application is lacking-only isolated retrospective studies have reported progestogen resistance or disease progression/recurrence in some patients. Preliminary data from our team showed that all 14 POLEmut EC patients receiving FST (including FIGO 2023 Stage IA2 G2, Stage IC G3, and progestogen-insensitive cases) achieved CR; an additional 6 POLEmut EC patients treated with ICIs also attained CR.

   Based on this evidence, this study proposes PD-1 monoclonal antibody monotherapy for POLEmut EC patients with strong fertility preservation demands, while expanding FST eligibility to FIGO 2023 Stage IA. The primary objectives are to evaluate FST efficacy, oncological outcomes, and reproductive outcomes of ICIs.
2. MMRd/MSI-H EC MMRd/MSI-H EC constitutes 25%-33% of all EC cases, featuring TMB-H (≥10 mutations/Mb), dense intratumoral CD8+ T cells, tertiary lymphoid structures, and high PD-1/PD-L1 expression. However, its response rate to progestogens is significantly lower than that of NSMP EC, with higher recurrence rates (potentially associated with activation of progesterone receptor-independent pathways). Currently, ICIs are approved for the treatment of pretreated advanced MMRd/MSI-H EC (objective response rate: 39%-49.1%, with durable efficacy and manageable toxicity). Early-phase clinical trials have further confirmed their potential: in a Phase II trial involving resectable Stage I-III MMRd solid tumors (including EC), 49 patients with MMRd locally advanced rectal cancer achieved clinical CR after 6 months of PD-1 inhibitor (dostarlimab) neoadjuvant therapy and avoided surgery; among 54 patients with non-rectal MMRd solid tumors, 35 achieved clinical CR (33 avoided surgery). Of 103 patients completing treatment across both cohorts, 84 achieved clinical CR (82 avoided surgery), with a 2-year RFS rate of 92% among 117 patients and 95% of adverse events being reversible Grade 1-2. In the EC-specific setting, 12 out of 15 patients with resectable Stage I-III MMRd/MSI-H EC achieved clinical CR after 6 cycles of nivolumab (480mg Q4W); 7 of these patients avoided surgery with no recurrence during follow-up (first enrollment: February 2019). Additionally, literature has reported successful pregnancy in a Lynch syndrome (MMRd-associated) patient after achieving CR with PD-1 monoclonal antibody; our team's preliminary data showed CR in all 4 Lynch syndrome patients (including those refractory to conventional progestogen therapy) treated with PD-1 monoclonal antibodies, suggesting ICIs may outperform progestogens.

   Notably, MMRd exhibits internal heterogeneity: based on genetic mechanisms, it can be classified into MLH1 promoter methylation subtype (poorer response to immunotherapy) and MMR gene mutation subtype (nearly 100% response rate to immunotherapy in patients with germline mutations, including Lynch and Lynch-like EC). Therefore, this study proposes an "ICI ± progestogen" regimen for MMRd EC patients undergoing FST: patients with confirmed germline or somatic MMR gene mutations will receive ICI monotherapy, while those with MLH1 methylation will receive ICI combined with high-dose potent progestogens. FST eligibility will be expanded to FIGO 2023 Stage II, with objectives to evaluate regimen efficacy, oncological/reproductive outcomes, and analyze efficacy differences and potential mechanisms across MMRd patients with distinct genetic backgrounds.
3. NSMP EC As the most common EC subtype (32%-49% of all cases), NSMP EC can be stratified into high-risk and low-risk groups based on ER expression. The low-risk subtype, predominantly ER-positive endometrioid carcinoma, represents the main population for FST, with high-dose progestogens as the standard regimen. Retrospective studies showed that NSMP EC patients undergoing FST achieved a 6-month CR rate and overall CR rate (72%, 18/25) significantly higher than ER/PR-positive MMRd patients (37.5%, 6/16) in the same period, with a lower recurrence rate (17.4% vs. 83.3%, p<0.05). However, clinically, 70%-80% of patients with early EC/atypical endometrial hyperplasia (AEH) require 9-10 months to achieve CR, and approximately 1/3 of patients either require over 9 months of treatment or remain non-responsive. Our team's preliminary research has identified PTEN mutation²⁷, SIGLEC10 mutation, insulin resistance, and obesity as key predictive factors for progestogen insensitivity, and established a progestogen sensitivity prediction model.

Simultaneously, our team discovered that progestogen-insensitive/refractory EC patients can still achieve CR with the "gonadotropin-releasing hormone agonist (GnRHa) combined with aromatase inhibitor (AI, mainly letrozole)" regimen. This regimen inhibits EC proliferation by suppressing estrogen production in the ovaries and peripheral tissues: GnRHa inhibits ovarian function and reduces estrogen levels within 14 days of administration, while letrozole blocks aromatase activity to inhibit the conversion of androstenedione to estrone/estradiol-representing a mechanism distinct from progestogens. Clinical studies have verified its feasibility: Zhang et al. reported a 100% CR rate (CR duration: 3-6 months) in 6 young obese EC patients treated with this regimen; Zhou et al. achieved CR rates of 88.2% (15/17) in early endometrioid EC (EEC) and 100% (12/12) in AEH patients using "GnRHa combined with LNG-IUS or letrozole" (median treatment duration: 18.7 months);A small-sample retro spective study showed that EEC/AEH patients achieving CR with this regimen had significantly longer disease-free survival than those treated with high-dose progestogens (hazard ratio: 2.158; 95% CI: 0.948-4.913). Additionally, this regimen avoids significant weight gain, causes minimal liver/kidney dysfunction, and prevents adverse events such as vaginal bleeding and breast cancer, thereby improving patient adherence. The ovarian protective effect of GnRHa may also enhance pregnancy rates after CR. However, attention should be paid to GnRHa-induced "medical ovarian ablation" complications (hot flashes, night sweats, osteoporosis) and the long-term hypoestrogenic effects of AIs on bone metabolism, which require close follow-up and timely intervention in the study.

Based on the above evidence, this study proposes progestogen sensitivity prediction model-guided stratified precision treatment for low-risk NSMP EC patients: patients predicted to be progestogen-sensitive will receive classical high-dose potent progestogens (MA/MPA), while those predicted to be progestogen-insensitive will receive "GnRHa combined with letrozole".

3 Research Objectives

To evaluate the FST efficacy and reproductive outcomes of different fertility-sparing regimens based on EC molecular subtypes. As the world's first prospective multicenter umbrella clinical trial optimizing EC FST protocols based on molecular characteristics, this study aims to:

1. Develop personalized FST regimens for POLEmut, MMRd/MSI-H, and NSMP EC subtypes-namely "ICI monotherapy", "ICI ± progestogen", and "progestogen sensitivity-stratified therapy"-to optimize existing FST strategies;
2. Expand FST eligibility to FIGO 2023 Stage IA for POLEmut EC and FIGO 2023 Stage II for MMRd/MSI-H EC, breaking the limitations of current indications;
3. Improve FST CR rate, shorten CR duration, reduce adverse events, and enhance patients' reproductive and oncological outcomes;
4. Explore and validate FST efficacy predictors and prognosis-related biomarkers for each subtype, improve the accuracy of disease risk control and prognostic assessment, and provide high-quality clinical evidence for optimizing EC FST protocols.

4 Research Methods Study Design: Prospective, open-label, multicenter, umbrella clinical trial Study Population: Patients with early-stage endometrial carcinoma requiring fertility-sparing treatment

This is a non-randomized controlled, prospective, multicenter, umbrella clinical trial implementing stratified management based on molecular subtypes:

1. POLEmut Stage II Single-Arm Interventional Study: Enroll patients with FIGO 2023 Stage IA POLE-mutant endometrial carcinoma to evaluate the CR rate, CR duration, and reproductive outcomes of ICI monotherapy in FST with expanded indications. Enrolled patients will receive ICI monotherapy.
2. MMRd Stage II Single-Arm Interventional Study: Stratify patients based on MLH1 methylation status/MMR coding gene mutation status. Patients with MMR coding gene mutations (somatic/germline) will receive ICI monotherapy; MMRd patients with MLH1 promoter methylation will receive ICI combined with high-dose potent progestogens (PD-1 + MPA/MA). The study will evaluate the CR rate, CR duration, and reproductive outcomes of FST with expanded indications.
3. NSMP Stage III Two-Arm Interventional Study: Based on the prediction model, progestogen-sensitive patients will receive high-dose potent progestogens (MA/MPA); progestogen-insensitive patients will receive "GnRHa combined with letrozole". The study will evaluate FST efficacy and reproductive outcomes while further validating the predictive value of the model.
4. exclusion from FST: NSMP EC with ER negativity and/or L1CAM positivity (≥10%) or p53abn endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 45 years;
2. Strong willingness to preserve fertility/uterus: Patients who have fertility requirements and insist on preserving fertility; or patients who have no fertility requirements but insist on preserving the uterus;
3. Newly diagnosed endometrial cancer: Pathologically diagnosed as endometrial cancer via endometrial biopsy, diagnostic dilation and curettage, or hysteroscopic examination;
4. Recurrent patients: Patients with endometrial lesions who received conservative treatment previously and developed recurrent endometrial cancer, with an interval of more than 6 months from the last standardized treatment, or deemed eligible for enrollment by the researcher after evaluation;
5. Imaging examinations (including pelvic enhanced MRI, upper abdominal enhanced CT/MRI, chest non-contrast CT, or PET/CT-MR) performed within 2 weeks before enrollment treatment initiation to confirm that the lesions are confined to the uterus without extrauterine involvement; for patients allergic to iodine contrast agents, MRI can be used instead of CT;
6. Clear molecular subtypes: POLE-mutant, NSMP (no specific molecular profile), or MSI-H (microsatellite instability-high);
7. Provide informed consent and sign the informed consent form;
8. Good compliance and follow-up conditions, willing and able to complete scheduled follow-up visits at our hospital;
9. No significant abnormalities in major organ functions, with relevant test values meeting the following requirements:White blood cell count ≥ 3×10⁹/L or absolute neutrophil count ≥ 1.5×10⁹/L; Platelet count ≥ 100×10⁹/L; AST and/or ALT < 2× upper limit of normal (ULN); Serum creatinine < 2× ULN;
10. Karnofsky Performance Status (KPS) score ≥ 90; Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
11. Concurrent use of thyroid medications, calcium tablets, vitamin D, bisphosphonates, metformin, aspirin, etc., is permitted;
12. Multidisciplinary Team (MDT) discussion is required before treatment initiation.
13. Additional Targeted Inclusion Criteria Based on Different Molecular Subtypes： 1) POLE-mutant endometrial cancer: Pathologically and radiologically evaluated as FIGO 2023 Stage IA endometrial cancer; 2). dMMR (deficient mismatch repair)/MSI-H endometrial cancer: Pathologically and radiologically evaluated as FIGO 2023 Stage I-II endometrial cancer; Patients with Lynch syndrome may have other Lynch-related tumors in other systems; 3) NSMP endometrial cancer: Pathologically and radiologically evaluated as FIGO 2023 Stage IA1 endometrioid carcinoma; Pathological grade: G1/G2; Lesions confined to the endometrial layer; Immunohistochemistry: ER-positive, L1CAM-negative (< 10% positive cells).

Exclusion Criteria:

1. Unclear molecular subtype or refusal to undergo molecular subtyping;
2. p53-abnormal molecular subtype;
3. ER-negative confirmed by pathological immunohistochemistry;
4. L1CAM-positive confirmed by pathological immunohistochemistry (L1CAM ≥ 10% positive cells);
5. Received any of the following treatments within 6 months before enrollment: high-dose potent progestins (megestrol acetate or medroxyprogesterone acetate) for consecutive ≥ 3 months; GnRHa ± letrozole for consecutive ≥ 3 months; immune checkpoint inhibitors for consecutive ≥ 3 months; levonorgestrel-releasing intrauterine system (Mirena) for consecutive ≥ 3 months; other treatments that may affect efficacy evaluation;
6. Contraindications to therapeutic drugs (immune checkpoint inhibitors, progestins, GnRHa, letrozole);
7. Complicated with severe medical diseases or severe liver dysfunction;
8. History of major organ transplantation;
9. History of severe mental illness or cerebral functional disorders;
10. History of autoimmune diseases requiring immunosuppressant therapy;
11. History of substance abuse or drug addiction;
12. Request for hysterectomy or other treatments except conservative drug therapy;
13. Inability to comply with the study protocol;
14. POLE-mutant/NSMP endometrial cancer: Complicated with other gynecological malignancies; For non-gynecological malignancies, enrollment is permitted if MDT evaluation confirms no impact on fertility-preserving treatment, and excluded if it affects fertility-preserving treatment or efficacy evaluation;
15. dMMR/MSI-H endometrial cancer (non-Lynch syndrome): Complicated with other malignancies, and MDT evaluation confirms impact on the selection of fertility-preserving treatment regimens or efficacy evaluation.

Exclusion Criteria for Immune Checkpoint Inhibitor Use:

1. Previous treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or drugs targeting other stimulatory or co-inhibitory T-cell receptors (e.g., CTLA-4, OX-40, CD137);
2. Received or planned to receive live vaccines within 30 days before the first dose of study intervention. Note: Inactivated vaccines are permitted;
3. Known intolerance to study interventions (or any excipients);
4. Diagnosed with immunodeficiency or receiving chronic systemic steroid therapy (≥ 10 mg prednisone per day or equivalent dose) or any other form of immunosuppressive therapy within 7 days before the first dose of study intervention;
5. Severe hypersensitivity reaction (≥ Grade 3) to PD-1/PD-L1 monoclonal antibodies and/or any of their excipients;
6. Active autoimmune diseases requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within the past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic treatment and is permitted;
7. History of (non-infectious) pneumonitis requiring steroid treatment or current pneumonitis;
8. Active infection requiring systemic treatment;
9. Known history of HIV infection;
10. Known history of hepatitis B (defined as HBsAg-positive) or active hepatitis C virus infection (defined as detectable HCV RNA [qualitative]); a. Chronic hepatitis B virus (HBV) carriers: HBV carriers with normal liver function and low HBV DNA load (e.g., below the lower limit of detection or at a low level) may be considered for PD-1 treatment after comprehensive evaluation. During PD-1 treatment, close monitoring is required, and appropriate antiviral prophylaxis should be administered if necessary to ensure treatment safety and efficacy; b. Patients with well-controlled hepatitis B: Patients with hepatitis B who have achieved good disease control through long-term standardized antiviral treatment, with mild liver inflammation and fibrosis, basically normal liver function, and no obvious complications such as cirrhosis or liver failure may receive PD-1 treatment;
11. Any history or current evidence of diseases, treatments, or laboratory abnormalities that the researcher believes may confound study results, interfere with the patient's ability to complete the study, or make trial participation not in the patient's best interest;
12. Known mental illness or substance abuse disorder that may interfere with the patient's ability to comply with study requirements;
13. Other exclusion criteria: Previous allogeneic tissue/solid organ transplantation; Failure to fully recover from surgery and/or any surgical complications;
14. Currently breastfeeding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The complete response rate (CRR) at 32 weeks after initiating treatment. | 32 full weeks following the first administration of fertility-preserving treatment for early-stage endometrial cancer patients.
  This endpoint aims to assess the therapeutic response of patients stratified by molecular subtypes ( POLE-mutant, MSI-H, and NSMP). The complete response rate (CRR) is defined as the proportion of patients in each molecular subtype cohort who achieve complete disappearance of all detectable endometrial lesions, confirmed by a combination of hysteroscopic examination and endometrial biopsy (pathologically negative for cancer cells).

SECONDARY OUTCOMES:
the complete response rate (CRR) at 16 weeks after initiating treatment. | 16 full weeks following the first administration of fertility-preserving treatment for early-stage endometrial cancer patients.
  This endpoint aims to assess the 16 weeks' response of patients stratified by molecular subtypes ( POLE-mutant, MSI-H, and NSMP). The complete response rate (CRR) is defined as the proportion of patients in each molecular subtype cohort who achieve complete disappearance of all detectable endometrial lesions, confirmed by a combination of hysteroscopic examination and endometrial biopsy (pathologically negative for cancer cells).
Median treatment duration to achieve complete response in study cohorts with different molecular subtypes | through study completion, an average of 1 year.
  The median duration is calculated using the Kaplan-Meier method, with the start time anchored to the first day of treatment and the end time marked as the date of the pathological report confirming complete response. Patients who do not achieve complete response by the end of the study (32 weeks) or who discontinue treatment early due to progression, adverse events, or personal reasons will be classified as "censored" in the statistical analysis, and their follow-up status will be clearly recorded.
Adverse Reactions and Safety Profiles of Different Fertility-Preserving Treatment Regimens | Throughout study completion, an average of 1year
  Safety is evaluated based on the incidence, severity, and resolution of adverse reactions (ARs) associated with each treatment regimen. ARs are graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, including grade 1 (mild) to grade 5 (death).
Impact of Different Treatment Regimens on Ovarian Function | at four time points: (1) Baseline (within 1 week before treatment initiation); (2) 16 weeks after treatment; (3) 32 weeks after treatment; (4) The time point of complete response (if achieved earlier than 32 weeks).
  Specific evaluation indicator: anti-Müllerian hormone (AMH) .The impact of treatment is defined as the relative change in AMH from baseline, with a focus on identifying whether the treatment causes reversible or irreversible damage to ovarian reserve.
Quality of Life of Patients Receiving Different Treatment Regimens | Assessments are conducted at the same four time points as ovarian function evaluation (baseline, through study completion, an average of 1year).
  Quality of life (QoL) is evaluated using validated international scales
Disease Recurrence Rate Within 2 Years After Achieving Complete Response During Follow-Up | The follow-up period starts from the date of confirmed complete response and lasts for 24 consecutive months.
  Recurrence is defined as the re-emergence of endometrial cancer lesions (confirmed by pathology), or the occurrence of extrauterine metastases (e.g., pelvic lymph node, ovarian, or distant organ metastases) confirmed by imaging (MRI/CT/PET-CT) and/or pathology.The recurrence rate is calculated as the number of patients with recurrence divided by the total number of patients who achieved complete response. For patients lost to follow-up, the last follow-up date is used as the censoring time, and the reason for loss to follow-up is recorded.
Pregnancy Rate within 2 Years After Achieving Complete Response During Follow-Up | starting from the date of complete response and ending at 2 years or the time of the first pregnancy (whichever comes first).
  This endpoint focuses on the reproductive potential of patients after successful fertility-preserving treatment, with follow-up starting from the date of complete response and ending at 2 years or the time of the first live birth (whichever comes first). Pregnancy rate: the proportion of patients who achieve clinical pregnancy (confirmed by ultrasound showing intrauterine gestational sac and fetal heartbeat) after natural conception or assisted reproductive technology (ART, e.g., in vitro fertilization-embryo transfer);
Live birth rate within 2 Years After Achieving Complete Response During Follow-Up | starting from the date of complete response and ending at 2 years or the time of the first live birth (whichever comes first).
  Live birth rate: the proportion of patients who deliver a viable infant (born after ≥24 weeks of gestation) among those who achieved clinical pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: XIAOJUN CHEN, PhD. MD., Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No